CLINICAL TRIAL: NCT04325477
Title: A Feasibility, Short-term Study With a Novel, Dynamic, and Disposable Over the Counter Device for Stress Urinary Incontinence
Brief Title: A Feasibility Study With a Novel, Dynamic and Disposable Over-the-counter Device for Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynamics LTD (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NLX-010
Record Dates: First submitted 2020-03-20; First posted 2020-03-27 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Stress Urinary Incontinence
Keywords: intravaginal device; pad weight gain; stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: A prospective one-arm study with subjects serving as their own control.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nolix Device (Experimental): Comparing use of device to non-treatment (pads only) phase
  Interventions: Device: Nolix Device

INTERVENTIONS:
Device: Nolix Device — The Nolix device is a single use, dynamic, and soft flexible intra-vaginal device for temporary management of SUI

SUMMARY:
This study was designed as an open label, feasibility, single-center, cross-over prospective study in women with stress urinary incontinence. Subjects served as their own control.

DETAILED DESCRIPTION:
The primary objectives of this feasibility study were to evaluate the short-term efficacy of the Nolix device by measuring a reduction of SUI following a modified 1-hour PWG test and to measure the safety of the Nolix device based on adverse events that were reported by subjects during the study. The secondary objective was to assess usability and patient satisfaction using the Nolix device.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 21 and above
* Suffering from Stress Urinary Incontinence
* Women who can understand the nature of the study, are physically able to perform all required tasks and consent to it by signing a written Informed Consent Form prior to participation in the study

Exclusion Criteria:

* Age ≤ 21 years
* Pregnant or planning to become pregnant during the study.
* Vaginal birth or Cesarean section for the last 3 months prior to entering the study.
* Severely atrophic vagina.
* A history of Toxic Shock Syndrome (TSS).
* Active urinary tract or vaginal infection.
* Patients prone to recurrent vaginal or urinary tract infections (i.e. more than 3 times in the past year).
* Has experienced unusual or unexpected vaginal bleeding within the last 6 months.
* Vaginal surgery within the last 3 months prior to entering the study.
* Has experienced difficulties with the use of intra-vaginal devices, including tampons.
* Presence of any condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Average daily PWG as measured in the baseline pad period is less than 4 grams /12 hours.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Continuous percent change in urine leakage | Pads were measured before and immediately after the 1 hour PWG test
  Continuous percent change in urine leakage is defined as: 100%*(PWG without Nolix - PWG with Nolix)/PWG without Nolix.
Change in the dryness of the pad | Pads were measured before and immediately after the 1 hour PWG
  Success ("1") if following the 1-hour PWG test, the pad weight increases by no more than 1 gram or Failure ("0") if following the 1-hour test, the pad weight increased by more than 1 gram.
Dichotomous change in urine leakage | Pads were measured before and immediately after the 1 hour PWG
  In accordance with FDA recommendations, the clinically meaningful level of improvement in PWG is at least 50%. Therefore, the dichotomous change is defined for each patient as follows: Success ("1"), if continuous percent change in PWG > 50% or Failure ("0"), if continuous percent change in PWG < 50%

SECONDARY OUTCOMES:
Comfort during Nolix use | 1 Day
  Comfort during Nolix device use will be measured through the Satisfaction Questionnaire, using a 10-point scale (where 1 is the most negative response and 10 the most positive, during the use of the device).
  Comfort during Nolix device use will be measured through the Benefit, Satisfaction, and Willingness to Continue Questionnaire, using a 10-point scale (where 1 is the most negative response and 10 the most positive, during the use of the device)
Overall satisfaction: Nolix Satisfaction Questionnaire | 1 Day
  Overall Satisfaction with the use of the Nolix device, as measured using the Nolix Satisfaction Questionnaire, selecting one of the following answers: 'Completely'; 'Somewhat'; or 'Not at all' (where 'Completely' is the most positive response and 'Not at all' is the most negative response).

CONTACTS AND LOCATIONS:
Overall Officials: Boris Friedman, Dr, Principal Investigator — Carmel Medical Center
Locations (1):
- Assuta Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
All personal data gathered in this trial will be treated in the strictest confidence by investigators, monitors, sponsor's personnel and independent ethics committee

REFERENCES:
- [Background] Krhut J, Zachoval R, Smith PP, Rosier PF, Valansky L, Martan A, Zvara P. Pad weight testing in the evaluation of urinary incontinence. Neurourol Urodyn. 2014 Jun;33(5):507-10. doi: 10.1002/nau.22436. Epub 2013 Jun 24. PMID 23797972
- [Derived] Naor MS, Kaploun A, Friedman B. A feasibility study with a novel, dynamic, and disposable over-the-counter device for the management of stress urinary incontinence. Neurourol Urodyn. 2021 Feb;40(2):653-658. doi: 10.1002/nau.24598. Epub 2020 Dec 21. PMID 33348425
- See also: Clinical Investigations of Devices Indicated for the Treatment of Urinary Incontinence - Guidance for Industry and FDA Staff — https://www.fda.gov/regulatory-information/search-fda-guidance-documents/clinical-investigations-devices-indicated-treatment-urinary-incontinence-guidance-industry-and-fda